CLINICAL TRIAL: NCT03962309
Title: Selection of People at Low Cardiovascular Risk: Development of an Inexpensive Pre-screening Algorithm Using Only Non-laboratory Measures. The SKIM Risk Study.
Acronym: SKIM
Status: Completed | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Centro Cardiologico Monzino (Other); IRCCS Multimedica (Other)
Responsible Party: Sponsor
Other Study IDs: IRFMN-7307
Record Dates: First submitted 2019-05-21; First posted 2019-05-24 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Epidemiology of Cardiovascular Risk
Keywords: Screening; General Practice; Self Assessment; Algorithms for risk stratification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients in charge of the participating GPs: In the study will be included patients in charge of the participating GPs aged 40-70 years
  Interventions: Other: Health self-assessment questionnaire

INTERVENTIONS:
Other: Health self-assessment questionnaire — The health self-assessment questionnaire includes questions covering anthropometric, sociodemographics, personal and family health history, life style habits and aspects of the behavioral domain. The questionnaire will be administered as paper format or web-based electronic format according to participants' preferences.

SUMMARY:
Early identification of individuals at high risk remains the cornerstone of primary cardiovascular prevention (CV). However, cardiovascular screening including people at low CV diseases (CVD) risk are too costly, time consuming and poorly effective in reducing incident CV events to be proposed at population level. Thus, innovative tools that allow to exclude low risk subjects in order to concentrate the relatively poor resources of NHS for primary prevention in high risk groups are needed. In this study, we will assess whether a new low cost strategy for CV risk stratification, based on non-laboratory measures, will allow to recognize low risk subjects who do not need further and expensive measures. To this end, we will take advantage of a General Practitioners (GPs) national network that will allow to work in the natural contest of primary prevention. If successful, the project will provide the basis for future, cost-effective prevention programs to be performed at national level.

DETAILED DESCRIPTION:
National, multicenter cross-sectional study.

The current study will be performed as part of Italian Cardiology Network implemented by the Italian Ministry of Health.

This study will be carried out with the collaboration with Study Center for Primary Care.

A random sample of subjects identified by the list of patients in charge of the participating GPs aged 40-70 years will be invited to a screening for the evaluation of their CV risk.

All patients who agree to participate in the study and sign the consent will complete a health self-assessment questionnaire which includes questions covering anthropometric, sociodemographics, personal and family health history, life style habits and aspects of the behavioral domain.

This will be followed by biometric measurements including height, weight and waist circumference conducted at the consulting room of the GP by certified staff. Informative predictors, selected among all variables selected, will be identified by a stepwise multivariable logistic regression. The low risk CV score will be calculated as the sum of the coefficients of the retained variables.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 40-70 years

Exclusion Criteria:

* Patients with previous cardiovascular events

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects aged 40-70 years in charge of GPs, giving the consent to partecipate in the study
Sampling Method: Non-Probability Sample
Enrollment: 2699 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
To develop of a low cost CVD risk score | 1 day
  The low cost CVD risk score will be developed using variable obtainable only by the self-assessment questionnaire (low-cost) to identify persons at low CVD risk according to Progetto CUORE or SCORE risk estimation.

SECONDARY OUTCOMES:
Race | 1 day
  Questions about the ethnic origin will be asked
Marital status | 1 day
  Questions about the marital status will be asked
Education status | 1 day
  Questions about the educational attainment will be asked
Employment status | 1 day
  Questions about the employment will be asked
Clinical Family History | 1 day
  Questions about the family health history will be asked
Personal Clinical History | 1 day
  Questions about the personal health history will be asked
The dietary habits | 1 day
  Questions about diet, alcohol consumption and salt consumption will be asked.
Physical activity | 1 day
  Questions about physical activity usually practiced will be asked
Smoking habits | 1 day
  Questions about smoking habits will be asked
Behavioral domain | 1 day
  Questions about aspects of the behavioral domain will be asked

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Latini, MD, Principal Investigator — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (3):
- Italy (3):
  - Cooperativa Medici Milano Centro, Milan
  - Cooperativa Nucleo Cure Primarie Val Pescara, Pescara
  - Cooperativa Medici 2000, Siena